CLINICAL TRIAL: NCT02160938
Title: Prenatal Cytogenetic Diagnosis by Array-Based Copy Number Analysis: Follow-Up
Brief Title: Prenatal Microarray Follow-Up Study
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Principal Investigator, Ronald J Wapner, MD, Professor and Vice Chairman for Research, Department of Obstetrics and Gynecology, Columbia University
Other Study IDs: AAAL0100; 5U01HD055651 (NIH)
Record Dates: First submitted 2014-06-10; First posted 2014-06-11 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Genetic Diseases
Keywords: microarray; prenatal; copy number variant; CNV; microdeletion; microduplication; genetic
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 3 year follow-up cohort: When the infants reach 24 months of age, the Study Follow-up Specialist will send all participants an age- appropriate Ages and Stages Questionnaire (ASQ) for completion.
  At as close to the age of 3 as possible, the following exams will be performed and are described below:
  * The Vineland-II Adaptive Behavior Scale (VABS)
  * Wechsler Preschool and Primary Scale of Intelligence IV (WPPSI-IV), or Wechsler Intelligence Scale for Children - Fifth Edition (WISC-V, for siblings older than 7 years 7 months, when necessary)
  * Children will also be photographed (for review by the study dysmorphologist)
  Interventions: Other: 3-year follow-up
- Limited follow-up cohort: Women with children who will not reach the age of 2 years 6 months by the end of our study but have a prenatally diagnosed CNV will be recruited into the limited follow-up study. Each center will describe the study to eligible women and will verbally obtain their permission to be contacted by the Study Follow-up Specialist. The Study Follow-Up Specialist will contact the patient, explain the study, and obtain full written informed consent.

INTERVENTIONS:
Other: 3-year follow-up — When the infants reach 24 months of age, the Study Follow-up Specialist will send all participants an age- appropriate Ages and Stages Questionnaire (ASQ) for completion.
  At the age of 3, the following exams will be performed and are described below:
  * The Vineland-II Adaptive Behavior Scale (VABS)
  * Wechsler Preschool and Primary Scale of Intelligence IV (WPPSI-IV), or Wechsler Intelligence Scale for Children - Fifth Edition (WISC-V, for siblings older than 7 years 7 months, when necessary)
  * Children will also be photographed (for review by the study dysmorphologist)
  Groups: 3 year follow-up cohort

SUMMARY:
The objectives of this multi-center collaborative study are to ascertain the frequency of specific copy number variants (CNVs) identified prenatally and to evaluate in detail through continued follow-up of the children the phenotypes associated with CNVs of known or uncertain clinical significance.

DETAILED DESCRIPTION:
Specifically the aims are as follows:

1. Determine the intellectual function of the children at age 3 years
2. Determine phenotypic characteristics other than intellectual function of the children at age 3 years
3. Determine the frequency of specific copy number variants discovered during routine prenatal diagnostic testing
4. Evaluate the educational, counseling and psychosocial implications of microarray testing as it is introduced as a standard prenatal diagnostic procedure.

ELIGIBILITY:
Eligibility Criteria for Enrollment into the 3 year Follow-up Cohort

Inclusion Criteria

1. Singleton or multi-fetal pregnancy with a prenatal invasive procedure resulting in a diagnosis by microarray analysis of a microdeletion/duplication less than 10 Mbs, either pathogenic or of uncertain significance, which is reported to the patient. This includes:

   * Infants diagnosed during prenatal diagnostic studies performed at the10 pre-specified prenatal diagnostic centers
   * Infants diagnosed by analysis of microarrays performed at the collaborating laboratories
   * Infants referred through the Prenatal Microarray Resource Center website
   * Children who will be at least 3 years of age by January of 2018, and who had a prenatally detected CNV <10 Mbs, either pathogenic or of uncertain significance OR
2. Children whose mothers were enrolled in the initial study (through July 2011) and who met inclusion criteria for follow-up in that phase, referred to as the "Index cohort". This includes:

   * CNVs of uncertain or known significance, some of which were not reported to the patient
   * Mosaic findings by karyotype and/or microarray alone.

Exclusion Criteria

1. Patient refusal to allow infant follow-up through the age of three
2. Patient not fluent in the English language
3. Patient under the age of 18
4. In surrogate pregnancies, the "rearing parents" are unavailable to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing prenatal microarray testing during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2013-02; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Full Scale Intelligence Quotient (IQ) score | age 3 years
  Full Scale IQ score from the Wechsler Preschool and Primary Scale of Intelligence IV or Wechsler Intelligence Scale for Children 5th edition

SECONDARY OUTCOMES:
Percent of subjects with specific commonly occurring CNVs | detected prenatally
Percent of subjects with seizure disorders | age: up to 3 years
Percent of subjects with cerebral palsy | age: up to 3 years
Percent of subjects with dysmorphic features diagnosed by dysmorphologist | age 3 years
Percent of subjects with structural anomalies | age: up to 3 years
Verbal Comprehension composite score | age: up to 3 years
  Verbal Comprehension composite score from the Wechsler Preschool and Primary Scale of Intelligence IV
Visual Spatial composite score | age: up to 3 years
  Visual Spatial composite score from the Wechsler Preschool and Primary Scale of Intelligence IV
Working Memory composite score | age: up to 3 years
  Working Memory composite score from the Wechsler Preschool and Primary Scale of Intelligence IV
Communication domain score | age: up to 3 years
  Communication domain score from the Vineland Adaptive Behavior Scale
Daily Living Skills domain score | age: up to 3 years
  Daily Living Skills domain score from the Vineland Adaptive Behavior Scale
Socialization domain score | age: up to 3 years
  Socialization domain score from the Vineland Adaptive Behavior Scale
Motor Skills domain score | age: up to 3 years
  Motor Skills domain score from the Vineland Adaptive Behavior Scale
Adaptive Behavior Composite score | age: up to 3 years
  Adaptive Behavior Composite score from the Vineland Adaptive Behavior Scale
Age-adjusted Z scores for birth weight | birth
Age-adjusted Z scores for birth length | birth
Age-adjusted Z scores for head circumference | birth

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Wapner, MD, Principal Investigator — Columbia University
Locations (9):
- United States (9):
  - Center for Fetal Medicine, Los Angeles, California
  - George Washington University Biostatistics Center, Rockville, Maryland
  - Montefiore Medical Center, Larchmont, New York
  - North Shore LIJ, Manhasset, New York
  - Mt. Sinai Medical Center, New York, New York
  - Columbia University, New York, New York
  - OB/GYN Services PC, New York, New York
  - Geisinger Health System, Danville, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Wapner RJ, Martin CL, Levy B, Ballif BC, Eng CM, Zachary JM, Savage M, Platt LD, Saltzman D, Grobman WA, Klugman S, Scholl T, Simpson JL, McCall K, Aggarwal VS, Bunke B, Nahum O, Patel A, Lamb AN, Thom EA, Beaudet AL, Ledbetter DH, Shaffer LG, Jackson L. Chromosomal microarray versus karyotyping for prenatal diagnosis. N Engl J Med. 2012 Dec 6;367(23):2175-84. doi: 10.1056/NEJMoa1203382. PMID 23215555
- [Background] Bernhardt BA, Soucier D, Hanson K, Savage MS, Jackson L, Wapner RJ. Women's experiences receiving abnormal prenatal chromosomal microarray testing results. Genet Med. 2013 Feb;15(2):139-45. doi: 10.1038/gim.2012.113. Epub 2012 Sep 6. PMID 22955112
- [Result] Bernhardt BA, Kellom K, Barbarese A, Faucett WA, Wapner RJ. An exploration of genetic counselors' needs and experiences with prenatal chromosomal microarray testing. J Genet Couns. 2014 Dec;23(6):938-47. doi: 10.1007/s10897-014-9702-y. Epub 2014 Feb 27. PMID 24569858